CLINICAL TRIAL: NCT06471387
Title: Exploring the Genetic and Molecular Underpinning of Nicotine Addiction for the Development of New Therapeutic Strategies
Brief Title: Unraveling the Genetic Basis of Nicotine Addiction for Novel Therapeutic Strategies
Acronym: NicoGen
Status: Recruiting | Type: Observational
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Panos Zanos, Assistant Professor, University of Cyprus
Other Study IDs: Onisilos2023; Onisilos-co-fund182 (Other Grant/Funding Number: Onisilos co-fund scheme)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Smoking Cessation; Smoking Cessation Intervention; Nicotine Addiction; Epigenetics; Molecular Biology; Genetic Epidemiology
Keywords: Nicotine Addiction; Smoking Cessation; Mendelian Randomization; Methylation; Genetic Epidemiology; Drug Repurposing; Epigenetic Biomarkers
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abstainers: Participants who achieve biochemically-verified smoking abstinence for at least 6 months following a cessation attempt aided by a computerized intervention program.
  Interventions: Behavioral: Flexiquit Smoking Cessation Intervention
- Relapsers: Participants who do not achieve abstinence and relapse to smoking following the cessation attempt.
  Interventions: Behavioral: Flexiquit Smoking Cessation Intervention

INTERVENTIONS:
Behavioral: Flexiquit Smoking Cessation Intervention — Participants will enter a 6-week (once weekly) self-delivered computerized intervention program called Flexiquit. Developed and validated by Clinical Psychologists of the Department of Psychology at the University of Cyprus, Flexiquit is an avatar-led app designed to support smoking cessation. It aims to assist with abstinence and monitor participants' progress through personalized modules and assessments.

SUMMARY:
This case-control study aims to investigate the genetic and molecular bases of nicotine addiction to identify potential therapeutic targets. The project will involve drug repurposing using Mendelian Randomization, a smoking cessation intervention, and the analysis of methylation status in participants undergoing nicotine withdrawal.

DETAILED DESCRIPTION:
Cigarette smoking remains the largest preventable risk factor for chronic diseases and premature mortality worldwide. While several medications have been approved to aid smoking cessation, most individuals relapse following an initial period of abstinence, with only around 15% achieving long-term abstinence beyond 6-12 months. This highlights a critical need to identify novel drug targets and develop more effective pharmacotherapies to treat nicotine addiction and maintain long-term smoking abstinence.

The proposed case-control study aims to leverage an interdisciplinary approach combining genetic epidemiology and molecular biology to: 1) Identify potential novel druggable targets for smoking cessation using a drug repurposing Mendelian randomization (MR) strategy, and 2) Assess whether epigenetic modifications (DNA methylation) of the identified drug target genes are associated with motivation to quit smoking, nicotine dependence severity, and vulnerability to smoking relapse following a cessation attempt.

Specifically, NicoGen study utilizes large-scale genomic datasets of expression quantitative trait loci (eQTLs) and protein quantitative trait loci (pQTLs) to identify genetic variants that influence expression/levels of genes encoding druggable proteins (targets of approved drugs/clinical candidates). MR analyses will then determine if genetically-predicted expression of these genes is causally related to smoking cessation outcomes.

Additionally, 200 current cigarette smokers (100 men, 100 women) will be recruited prior to smoking cessation for collection of biofluids for DNA extraction.

The methylation levels of the top candidate drug target genes identified in will be assessed and compared between: 1) Cases who achieve ≥6 month abstinence vs. relapsed controls, 2) High vs. low motivation to quit groups, and 3) High vs. low nicotine dependence groups. This allows identification of epigenetic biomarkers predictive of cessation outcomes.

Additionally, potential gender differences in the associations between gene methylation, motivation, dependence and relapse vulnerability will be explored to identify gender-specific drug targets.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years old
* Current daily cigarette smoker
* Able to understand study procedures and provide informed consent
* For females, non-pregnant and non-lactating

Exclusion Criteria:

* Presence of significant uncontrolled medical conditions (e.g. cardiovascular disease, respiratory disorders, cancer) that could affect smoking behaviors or study participation
* Presence of major uncontrolled psychiatric disorders (e.g. schizophrenia, bipolar disorder, severe depression)
* Current substance use disorder (except nicotine dependence)
* Taking medications that could significantly interfere with study objectives (e.g. medications for smoking cessation)
* Significant cognitive impairment that precludes ability to complete study procedures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of adult daily cigarette smokers recruited from communities across Cyprus who are able to attend study visits at the research facilities in Nicosia. Recruitment will leverage multiple avenues including primary care clinics, community outreach, word-of-mouth referrals, and smoking cessation services throughout the island. The goal is to enroll approximately 200 eligible participants, with equal representation of men and women, from both urban and rural areas of Cyprus. No other specific characteristics beyond meeting eligibility criteria are used to identify or restrict the source population.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Novel druggable gene targets for smoking cessation | Upon completion of Mendelian randomization analysis
  Genes encoding druggable proteins (targets of approved drugs or clinical candidates) whose genetically predicted expression levels are found to be causally associated with smoking cessation outcomes using Mendelian randomization approaches.
Association between methylation of candidate genes and nicotine dependence scores | Baseline
  Difference in methylation levels of top genes between participants with high vs. low scores on the Fagerström Test for Nicotine Dependence.
Association between DNA methylation of candidate drug target genes and motivation to quit smoking scores | 3 and 6 months post nicotine cessation
  Difference in methylation levels of the top candidate drug target genes between participants with high vs. low scores on a validated motivation to quit smoking questionnaire.
Association between methylation and smoking relapse vulnerability | 3 and 6 months post nicotine cessation
  Difference in methylation of top genes between cases achieving 6+ month abstinence vs. controls who relapsed to smoking.

SECONDARY OUTCOMES:
Gender differences in methylation associations | 3 and 6 months post nicotine cessation
  Differences between males and females in the associations between methylation of candidate genes and the motivation, dependence and relapse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Applied Neuroscience (CAN), Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karekla M, Savvides SN, Gloster A. An Avatar-Led Intervention Promotes Smoking Cessation in Young Adults: A Pilot Randomized Clinical Trial. Ann Behav Med. 2020 Oct 1;54(10):747-760. doi: 10.1093/abm/kaaa013. PMID 32383736